CLINICAL TRIAL: NCT01799460
Title: Mechanism Research of Traditional Chinese Medicine (the Comprehensive Treatment Regimen) in Treating Idiopathic Membranous Nephropathy by Genomewide Association Studies
Brief Title: Study on Single-nucleotide-polymorphism in Idiopathic Membranous Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiMEC-2011; 11YZ65 (Other Grant/Funding Number: Shanghai Municipal Education Commission)
Record Dates: First submitted 2013-01-08; First posted 2013-02-26 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: single-nucleotide-polymorphism; Traditional Chinese Medicine; the Comprehensive Treatment Regimen
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Glucocorticoids; Cyclosporine; Cyclophosphamide; Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CR/CTR group: The complete remission group treated by the Comprehensive Treatment Regimen
  Interventions: Drug: The Comprehensive Treatment Regimen of Traditional Chinese Medicine
- NR/CTR group: The non-remission group treated by the Comprehensive Treatment Regimen
  Interventions: Drug: The Comprehensive Treatment Regimen of Traditional Chinese Medicine
- CR/IA group: The complete remission group treated by Immunosuppressive Agents
  Interventions: Drug: The immunosuppressive agents
- NR/IA group: The non-remission group treated by Immunosuppressive Agents.
  Interventions: Drug: The immunosuppressive agents

INTERVENTIONS:
Drug: The Comprehensive Treatment Regimen of Traditional Chinese Medicine — ①ShenQiMoShen Decoction: which plays vital therapeutic effect in the CTR,the dosage is 150ml per serving and two services per day.Dosage and administration:150ml per time,twice per day
  ②HuoXueTongMai Capsule : which plays a vital role of promoting blood circulation and removing blood stasis. Its main components are the leeches. Dosage and administration: 4 capsules 3 times daily.
  ③HeiLiaoDou Particle: which will be prescribed when hypoproteinemia (serum albumin concentration≤30g/L)occurred and should be stopped taking until the serum albumin is above 30g/L. Dosage and administration: 2 packages 3 times daily.
  Other Names: ShenQiMoShen Decoction; HuoXueTongMai Capsule; HeiLiaoDou Particle
  Groups: CR/CTR group; NR/CTR group
Drug: The immunosuppressive agents — According to Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guideline for glomerulonephritis
  Other Names: Glucocorticoid; Cyclosporine; Cyclophosphamide; Tacrolimus
  Groups: CR/IA group; NR/IA group

SUMMARY:
The purpose of this study is to analysis the different genotype in the idiopathic membranous nephropathy patients which with different therapeutic outcomes after treated by the Comprehensive Treatment Regimen or immunosuppressive agents, and so as to looking for ideal markers to assess appropriate treatment approach and the long-term efficacy.

DETAILED DESCRIPTION:
The primary objective of this study is to looking for the gene level predictors in the patients who suffered from idiopathic membranous nephropathy. And according to the predictors, the clinicians could make a decision which method should be taken on IMN patients, Traditional Chinese Medicine or western medicine, and could get better results.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic membranous nephropathy
* Chronic Kidney Disease (CKD)≤3 stage（Glomerular Filtration Rate (GFR)≥30ml/min）and 24 hour urinary protein≥3g
* Voluntarily participated in the study and signed an informed consent

Exclusion Criteria:

* Combined life-threatening complications such as serious infection
* Abnormal glucose metabolism
* Patients with malignant tumors or malignancy , HIV infection and a history of mental illness , acute central nervous system disease , serious gastrointestinal diseases,etc
* Pregnancy or breast-feeding women
* Undergoing other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: idiopathic membranous nephropathy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Genome-wide single-nucleotide-polymorphism of IMN patients treated by the Comprehensive Treatment Regimen or conventional approach | one year
  Screening for single-nucleotide-polymorphism as the prognostic factor for the TCM intervention of IMN patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Lin, PHD,MD, Study Director — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China